CLINICAL TRIAL: NCT04906642
Title: Clinical Assessment of How Next Science XPERIENCE No Rinse Antimicrobial Solution May Promote Wound Healing by Decreasing Post-Operative Infections in Gustilo and Anderson Type II and IIIA or IIIB Tibial Fractures
Brief Title: Clinical Assessment of Next Science Solution on Gustilo and Anderson Type II and IIIA or IIIB Tibial Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low patient enrollment, less-than-ideal patient sample for the study, leading to a significant number of missed scheduled study visits, inefficient study data, and reallocation of finances.
Sponsor: Next Science TM (Industry)
Collaborators: Piedmont Healthcare (Other); Hughston Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSP-018
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Surgical Wound Infection
Keywords: Open tibial fracture; Surgical Site Infection; Surgical Irrigation; Single Stage Closure
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, double-blinded clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the double-blinded nature of the study, neither the participant, treating physician, site staff, or site study team will be aware of the treatment assignment (XPERIENCE No-Rinse Antimicrobial Solution or blinded saline) of each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Each of the following procedures will be conducted according to general or local site Standard of Care (SoC):
  * Medication administration at surgery
  * Surgical irrigation and wound debridement
  * Surgical fracture preparation/fixation
  * Surgical closure
  Interventions: Other: Standard of Care
- Standard of Care plus Next Science (Experimental): In addition to the SoC, the blinded product will be applied in place of saline irrigation as the wound is closed (after bone fracture preparation/fixation), depending on the randomization.
  Interventions: Device: Next Science

INTERVENTIONS:
Device: Next Science — Solution is a clear, colorless, aqueous solution that is used to remove debris, including microorganisms, from wounds via hydrodynamic shear across the wound. This aids in the removal of foreign material such as, microorganisms, dirt, and debris.
  Arms: Standard of Care plus Next Science
Other: Standard of Care — Normal Saline will be used in place of Next Science for irrigation
  Arms: Standard of Care

SUMMARY:
This is a prospective, randomized, controlled, double-blinded clinical feasibility study of subjects that are being treated for Gustilo and Anderson Type II or IIIA or IIIB Tibial Fractures

DETAILED DESCRIPTION:
This is a prospective, controlled, double-arm, double-blinded, randomized clinical study of 30 subjects that are undergoing single stage surgical repair of Type II or IIIA or IIIB tibial fractures.

Institutional Review Board (IRB) approval is required before the site can begin enrolling patients. Additionally, protocol amendments need to be approved by the IRB prior to starting any changes or procedures stemming from the amended protocol. Potentially eligible patients will be offered study enrollment and all subjects are required to participate in the informed consent process and sign the most recent IRB-approved written informed consent document prior to being enrolled in the study. If all the study inclusion/exclusion criteria are met, patients will be presented with the option to participate in the study and informed consent procedures will be carried out, in compliance with currently applicable subjects' rights and safety regulations. Reconsenting procedures for cases of protocol amendments will be performed in compliance with the IRB.

Patients who present for open tibial fracture repair surgery will have a pre-op medical evaluation prior to being screened against the protocol's inclusion/exclusion criteria. If criteria are met, patients will be presented with the option to participate in the study, and informed consent procedures will be carried out, in compliance with currently applicable participants' rights and safety regulations. At the time of surgery, participants determined to require surgical repair of a Type IIIC tibial fracture will be excluded. Patients who continue to be eligible meeting inclusion/exclusion criteria at the time of surgery will be randomized to one of the two treatment arms: SOC with Saline or SOC plus Next Science treatment. The treatment assignment will be predetermined by a randomization plan within Castor Electronic Data Capture (EDC) system. Although, paper source documents will be used to obtain subject data, randomization will be primarily through the EDC system. As a back-up, should the EDC system be unavailable at that time, randomization will occur using a sealed envelope system.

The following must have occurred prior to determining treatment assignment:

* Screening
* Participant must meet all eligibility requirements
* Informed Consent must be signed
* Continued Eligibility screening
* Randomization must occur*

  * Randomization occurs prior to surgery based on Exclusion #8. If the index fractures are bilateral, right leg will be randomized while the other leg will be assigned to the opposite treatment arm to prevent dosing of identical products on one subject.

Once surgical evaluation occurs if the index fracture is determined to be Type II, IIIA or IIIB (that does not require referral to another surgical service [vascular, plastic surgery] ) then the subject will continue to dosing. If the index fracture(s) must receive additional surgical referrals they will not be dosed, considered a screen failure, and exited from the study.

If the patient fails to meet continued eligibility:

* Screen Failure and
* Study Exit forms must be completed.

Accurate recording of the information per section 9.3 is critical for the traceability of treatment and product to a participant.

The duration of each subjects' participation once eligible and approved to start treatment, will start from Day 1 (first index surgery) and end at the Day 90 Visit. On-site visits will be carried out at Screening/Enrollment; Day of Surgery; Day of Discharge; and Days 14, 30, and 90; consisting of safety, bone healing (via X-ray findings), bioburden assessment, and surgical site infection assessment questions.

The key parameters of the study include bioburden and surgical site infection assessment, re-admission assessment, serious adverse events, and healthcare cost impact.

Bacterial identification and quantification will be evaluated via two methods: PCR/NGS (according to this protocol) and microbiology/pathology (according to site SOC). PCR/NGS swabs will be taken after fracture fixation inside the wound and then around the closed surgical incision:

* After fracture fixation (deep tissue): Swabs will be performed right after fracture fixation, before blinded rinse, and then immediately after blinded irrigation. The swabs will be performed on the entire wound base and around the fixation device. The time of collection for each swab must be specific (hour and minute) and recorded on the specimen label and requisition form.
* After closed surgical incision (superficial): After final closure, swabs will be taken within the 1-2cm perimeter surrounding the entire incision. This will be repeated on the day of discharge. The time of collection for each swab must be specific (hour and minute) and recorded on the specimen label and requisition form.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years old
2. Scheduled to undergo surgery to repair open tibial fracture
3. Willing and able to comply with all study procedures and be available for the duration of the study
4. Provide signed and dated informed consent or obtain consent from legally authorized representative
5. Not be pregnant, planning to become pregnant, or nursing female subjects.

Exclusion Criteria:

1. Unable to provide signed and dated informed consent or unable to obtain consent from a legally authorized representative
2. Unable or unwilling to comply with all study-related procedures
3. Known history of allergic reaction to any of the study products or its components, including any products used for standard of care (such as dressings or any coverings)
4. Subject has known history of contraindications to general anesthesia
5. Subject with any underlying condition or state that, in the investigator's opinion, will make them too critically ill to complete 30 and/or 90 day follow ups
6. Pregnant, planning to become pregnant, or nursing female subjects.
7. Any subject positive for Covid-19 virus at time of surgical screening
8. Tibial plateau, pilon, or Gustilo-Anderson type IIIc fractures and any fracture that will require referral to another surgical service will be excluded from this study
9. Any patient who will require ongoing use of NPWT after hospital discharge will be excluded from the study.
10. Subjects have evidence of prolonged QT segment, per EKG.
11. Subjects from a vulnerable population, in accordance with 45 CFR 46 Subparts B, C, and D

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | 90 days
  Proportion of subjects that develop a surgical site infection (superficial, deep, or organ space) from surgery to post-op Day 90 for the Next Science Group compared to the Control group.

SECONDARY OUTCOMES:
Superficial Bioburden | 90 days
  Mean change in bioburden around the closed incision, as evaluated via PCR/NGS, from baseline to Day of Discharge for the Next Science Group compared to the Control group.
Deep Bioburden | 1 day
  Mean change in bioburden from the deep tissue immediately after fixation around the fixation site, as evaluated via PCR/NGS, before and after use of the blinded product for the Next Science Group compared to the Control group

CONTACTS AND LOCATIONS:
Overall Officials: Robert Harris, MD, Principal Investigator — Piedmont Healthcare
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Piedmont Healthcare, Columbus, Georgia

IPD SHARING:
Plan to Share IPD: No